CLINICAL TRIAL: NCT03309514
Title: Clinical Investigation of Transplantation of Neural Stem Cell-derived Neurons for the Treatment of Parkinson's Disease
Brief Title: Transplantation of Neural Stem Cell-Derived Neurons for Parkinson's Disease
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: NeuroGeneration (Industry)
Responsible Party: Principal Investigator, Michel F. Levesque, MD, Principal Investigator, NeuroGeneration
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGN-9076
Record Dates: First submitted 2017-10-10; First posted 2017-10-13 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Biological: Intracerebral microinjections

INTERVENTIONS:
Biological: Intracerebral microinjections — Stereotactic delivery of cell suspension into basal ganglia structures

SUMMARY:
This is a prospective study to demonstrate the safety and efficacy of differentiated neurons-derived from adult CNS progenitors cells transplanted in selected patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give informed consent prior to study
2. Male or Female with Diagnostic Criteria of Parkinson's disease
3. Age 35 to 85 years old
4. Parkinson's disease not due to trauma, infection, brain tumor, cerebrovascular disease
5. Hoehn and Yahr Stage III or IV
6. Parkinson's disease observed in the absence of:

   * Oculomotor palsy
   * Cerebellar sign
   * Orthostatic hypotension (drop greater than 20mmHg in mean pressure)
   * Pyramidal sign
   * Amyotrophy
7. Good general health or stable medical condition well controlled, without contraindications to anesthesia

Exclusion Criteria:

1. Patients with severe dementia and brain atrophy on MRI
2. Patients with severe hypertension; renal, liver, cardiac or other major organ disease; coagulopathy; cancer; other significant systemic illnesses; hepatitis, HIV
3. Patients older than 85 or younger than 35
4. Patients who withhold informed consent
5. Patients with a history of alcohol or drug abuse
6. Sexually active women of childbearing potential without adequate form of birth control
7. Evidence of abnormal coagulation or anticoagulant therapy
8. Pregnancy or lactation
9. History of seizure disorders or current use of antiepileptic medication
10. Severe cognitive impairment
11. Clinically significant laboratory abnormality

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Motor UPDRS | 6 months
  UPDRS Motor scale